CLINICAL TRIAL: NCT01554748
Title: Improvement of Implant Survival in Total Joint Arthroplasty of the Trapeziometacarpal Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Torben B. Hansen, Professor, MD, PhD, Regional Hospital Holstebro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-01
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis
Keywords: total joint arthroplasty; thumb; trapeziometacarpal joint; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement

STUDY DESIGN:
Intervention Model Description: Implantation of TMC total joint arthroplasty in a patient cohort
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient cohort (Other): TMC total joint arthroplasty
  Interventions: Procedure: Total joint arthroplasty

INTERVENTIONS:
Procedure: Total joint arthroplasty

SUMMARY:
The study evaluates implant survival in total joint arthroplasty of the Trapeziometacarpal (TMC) joint by monitoring the survival of different implant types using radiostereometry (RSA) evaluation of the implants.

DETAILED DESCRIPTION:
The study evaluates implant survival and clinical outcome in total joint arthroplasty of the TMC joint. Different implant designs are included in the study both cemented and uncemented implants. Also the influence of patient factors and surgical technique on implant survival is investigated. The primary outcome is implant migration and loosening. Evaluation is done by monitoring migration and loosening of different implant types using RSA evaluation of the implants. Secondary outcomes are patient reported function evaluated with the Disability of the arm, shoulder and hand score (DASH) and visual analog pain score (VAS). Tertiary outcome is range of movement (ROM) plus grip strength.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Eaton type 2+3 TMC osteoarthritis

Exclusion Criteria:

* Patients with Eaton type 4 TMC osteoarthritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-01; Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 10 year survival
  Revision with removal of implant

CONTACTS AND LOCATIONS:
Overall Officials: Torben B. Hansen, MD, PhD, Principal Investigator — Orthopaedic Research Unit Regional Hospital Holstebro
Locations (1):
- Department of Orthopaedics, Regional Hospital Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Mosegaard SB, Stilling M, Hansen TB. Risk factors for limited improvement after total trapeziometacarpal joint arthroplasty. Health Qual Life Outcomes. 2020 Mar 30;18(1):90. doi: 10.1186/s12955-020-01333-z. PMID 32228611